CLINICAL TRIAL: NCT06052033
Title: The Effect of 5-aminolaevulinic Acid Photodynamic Therapy Versus C02 Laser in the Treatment of Persistent Cervical Low-grade Squamous Intraepithelial Lesions With High-risk HPV Infection:A Non-randomized Controlled Trail Study
Brief Title: Comparison of 5-ALA Photodynamic Therapy and CO2 Laser for Treating Persistent Low-Grade Cervical Lesions With High-Risk HPV Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, YANHU, director, First Affiliated Hospital of Wenzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2023-188
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: HPV-Related Cervical Carcinoma; Low-Grade Squamous Intraepithelial Lesions; HPV Infection; Photodynamic Therapy
Keywords: high-risk hpv infection; hpv persistent; Lsil; cervical lesions
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALA-PDT Group (Experimental): PDT involves cervical gel application and 25-minute laser light exposure. The procedure is repeated three times.
  Interventions: Procedure: CO2
- CO2 Laser Group (Other): CO2 laser therapy ablates cervical lesions with a depth of 7-10mm and a width of 3-5mm in a single session.
  Interventions: Procedure: CO2

INTERVENTIONS:
Procedure: CO2 — CO2 laser treatment is a surgical procedure that employs a high-powered carbon dioxide laser beam to precisely ablate cervical lesions. The laser is applied with a depth of 7-10mm and a width of 3-5mm beyond the lesion area in a single session. This intervention aims to address persistent low-grade cervical lesions associated with high-risk HPV infection.

SUMMARY:
Non-RCT clinical trial comparing 5-ALA photodynamic therapy and CO2 laser for persistent high-risk HPV-related low-grade cervical lesions.

DETAILED DESCRIPTION:
This non-randomized controlled trial aims to compare the effectiveness of two treatments, 5-aminolevulinic acid (5-ALA) photodynamic therapy and CO2 laser, for women with persistent low-grade cervical lesions associated with high-risk HPV infection lasting more than one year. The study's primary objective is to assess which treatment option yields better results. Participants in both groups will undergo specific therapeutic procedures, including 5-ALA photodynamic therapy or CO2 laser treatment. The study will analyze and compare the effects of these therapies on the regression or elimination of cervical lesions, offering valuable insights into the management of persistent low-grade cervical lesions among high-risk HPV-infected women.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years old with a history of sexual activity.
2. Subclinical infected individuals who have been confirmed as HR-HPV positive (if there is the same positive type in the typing test) for more than 1 year using HPV typing test, HPV E6/E7 mRNA test, HPV DNA test, and cervical triple step diagnostic procedure (cytology colposcopy histopathology).
3. Patients diagnosed with LSIL by pathological examination of cervical biopsy under colposcopy with an interval of more than 1 year.
4. No fundamental diseases of important organs.
5. Agree to receive treatment and/or follow-up according to regulations and sign an informed consent form.
6. There has been no history of using other drugs related to HPV infection in the past 3 months.

Exclusion Criteria:

1. HR-HPV persistent infection.
2. A total hysterectomy has been performed.
3. Concomitant endometrial cancer, ovarian cancer, and other reproductive tract tumors.
4. Complicated with abnormal heart, liver, and kidney functions, immune dysfunction, or immune system diseases such as systemic lupus erythematosus (SLE).
5. Using drugs such as immunosuppressants, antiviral agents, and glucocorticoids.
6. Pregnant and lactating women.
7. Acute reproductive tract inflammation.
8. Diabetes patients with uncontrolled blood sugar.
9. Patients who do not receive full treatment and follow-up.
10. Those who fail to sign the informed consent form.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Regression of Cervical Lesions. | Assessed at 6 months after the last PDT session.
  Measure the rate of regression in cervical lesions after three PDT sessions.

SECONDARY OUTCOMES:
Adverse Events. | Evaluated at 6 months after the CO2 laser treatment.
  Monitor and document any adverse events or complications related to CO2 laser treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- first affiliated hospital of Wenzhou medical university, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Wang Y, Xue J, Dai X, Chen L, Li J, Wu Y, Hu Y. Distribution and role of high-risk human papillomavirus genotypes in women with cervical intraepithelial neoplasia: A retrospective analysis from Wenzhou, southeast China. Cancer Med. 2018 Jul;7(7):3492-3500. doi: 10.1002/cam4.1559. Epub 2018 May 30. PMID 29851256
- [Result] Yang Y, Meng YL, Duan SM, Zhan SB, Guan RL, Yue TF, Kong LH, Zhou L, Deng LH, Huang C, Wang S, Wang GY, Wu DF, Zhang CF, Chen F. REBACIN(R) as a noninvasive clinical intervention for high-risk human papillomavirus persistent infection. Int J Cancer. 2019 Nov 15;145(10):2712-2719. doi: 10.1002/ijc.32344. Epub 2019 Apr 29. PMID 30989655
- [Result] Crosbie EJ, Einstein MH, Franceschi S, Kitchener HC. Human papillomavirus and cervical cancer. Lancet. 2013 Sep 7;382(9895):889-99. doi: 10.1016/S0140-6736(13)60022-7. Epub 2013 Apr 23. PMID 23618600
- [Result] Fu Y, Bao Y, Hui Y, Gao X, Yang M, Chang J. Topical photodynamic therapy with 5-aminolevulinic acid for cervical high-risk HPV infection. Photodiagnosis Photodyn Ther. 2016 Mar;13:29-33. doi: 10.1016/j.pdpdt.2015.12.004. Epub 2015 Dec 10. PMID 26687616
- [Result] Bhowmick R, Girotti AW. Signaling events in apoptotic photokilling of 5-aminolevulinic acid-treated tumor cells: inhibitory effects of nitric oxide. Free Radic Biol Med. 2009 Sep 15;47(6):731-40. doi: 10.1016/j.freeradbiomed.2009.06.009. Epub 2009 Jun 11. PMID 19524035
- [Result] Hu Z, Li J, Liu H, Liu L, Jiang L, Zeng K. Treatment of latent or subclinical Genital HPV Infection with 5-aminolevulinic acid-based photodynamic therapy. Photodiagnosis Photodyn Ther. 2018 Sep;23:362-364. doi: 10.1016/j.pdpdt.2018.07.014. Epub 2018 Jul 23. PMID 30048762
- [Result] Li D, Zhang F, Shi L, Lin L, Cai Q, Xu Y. Treatment of HPV Infection-Associated Low Grade Cervical Intraepithelial Neoplasia with 5-Aminolevulinic Acid-Mediated Photodynamic Therapy. Photodiagnosis Photodyn Ther. 2020 Dec;32:101974. doi: 10.1016/j.pdpdt.2020.101974. Epub 2020 Aug 21. PMID 32835877
- [Result] Wang X, You L, Zhang W, Ma Y, Tang Y, Xu W. Evaluation of 5-aminolevulinic acid-mediated photodynamic therapy on cervical low-grade squamous intraepithelial lesions with high-risk HPV infection. Photodiagnosis Photodyn Ther. 2022 Jun;38:102807. doi: 10.1016/j.pdpdt.2022.102807. Epub 2022 Mar 11. PMID 35288319
- [Result] Navarro Santana B, Sanz Baro R, Orozco R, Plaza Arranz J. Cervical vaporization in LSIL and persistent HPV infection. Taiwan J Obstet Gynecol. 2018 Aug;57(4):475-478. doi: 10.1016/j.tjog.2018.06.010. PMID 30122563